CLINICAL TRIAL: NCT01915836
Title: Quit IT: Development of a Web-based, 3D Coping Skills Game to Increase Self-Efficacy for Maintaining Smoking Abstinence Following Hospitalization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Muzzy Lane Software (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 11-043
Record Dates: First submitted 2013-08-01; First posted 2013-08-05 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Tobacco Use Cessation
Keywords: 11-043; MSKCC Tobacco Cessation Program
MeSH Terms: conditions — Tobacco Use Cessation | interventions — Surveys and Questionnaires

ARMS (1):
- Alpha game testers and questionaires (Experimental): This a video game designed to help smokers quit & remain non-smokers. Before the start the game,the participant will fill out a brief questionnaire.
  It should take about 5 minutes to complete. Once this is done, the game play should last about 30 minutes & will present with different scenes. These scenes will show situations that may trigger smoking urges such as walking into a room where another person is smoking. In the game, the participant will be able to use different ways of coping with urges to smoke such as taking several deep breaths or listening to music. The participant will be asked to talk aloud about what they think of the game. The participant will be video &/or audio recorded while doing this. Once finished testing the game, we will then ask you a few questions about what you thought of the game. We will also ask you how relevant different situations are to you as a smoker or someone who is trying to avoid smoking. The entire visit is expected to last about 1.5 hours.
  Interventions: Other: web-based video game (Quit IT); Behavioral: Questionnaires; Behavioral: Evaluation Interview

INTERVENTIONS:
Other: web-based video game (Quit IT)
Behavioral: Questionnaires
Behavioral: Evaluation Interview

SUMMARY:
The purpose of this study is to test a web-based video game to help cancer patients quit smoking. The investigators are interested in what participants like and do not like about the game.

ELIGIBILITY:
Inclusion Criteria:

* Treated by the MSKCC Tobacco Cessation Program
* At least 30 years of age

Exclusion Criteria:

* Insufficient manual dexterity and vision to use a computer and mouse as per self-report
* Unstable medical or psychiatric condition as determined by the PI and Co-PI.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-03; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Usability (10-item Game Usability Scale) | 1 time
  we will ask each participant to complete a Game Usability Scale3 which is a robust and highly recommended 10-item measure of usability developed for software testing that provides a global view of subjective assessments of usability.
Satisfaction | 1 time
  (users' subjective reactions to using the system) After the game play session, we will have participants complete an Avatar and Situation Menu Questionnaire so that participants can give feedback on 3 different avatars and 15 different coping with smoking challenges regarding how relevant each is to them as a smoker or someone trying to avoid smoking.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Ostroff, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Krebs P, Burkhalter J, Fiske J, Snow H, Schofield E, Iocolano M, Borderud S, Ostroff JS. The QuitIT Coping Skills Game for Promoting Tobacco Cessation Among Smokers Diagnosed With Cancer: Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Jan 10;7(1):e10071. doi: 10.2196/10071. PMID 30632971
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/